CLINICAL TRIAL: NCT04050540
Title: PrEP and dPEP: Doxycycline Post-exposure Prophylaxis for Prevention of Sexually Transmitted Infections Among Kenyan Women Using HIV Pre-exposure Prophylaxis
Brief Title: Doxycycline PEP for Prevention of Sexually Transmitted Infections Among Kenyan Women Using HIV PrEP
Acronym: dPEP-KE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); Kenya National AIDS & STI Control Programme (Other); University of California, San Francisco (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jared Baeten, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007487; R01AI145971 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections; HIV/AIDS; Neisseria Gonorrheae Infection; Chlamydia Trachomatis Infection; Syphilis Infection
Keywords: Sexually Transmitted Infections
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Gonorrhea; Sexually Transmitted Diseases | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dPEP Intervention Arm (Experimental): Participants assigned to dPEP will be instructed to take doxycycline 200 mg (two 100mg capsules) orally within 24 hours and up to 72 hours after each condomless sex act
  Interventions: Drug: Doxycycline
- Standard of Care Arm (No Intervention): Participants assigned to Standard of Care

INTERVENTIONS:
Drug: Doxycycline — 200 mg of doxycycline to be taken orally within 24 hours and up to 72 hours after each condomless sex act
  Arms: dPEP Intervention Arm

SUMMARY:
This is a randomized clinical trial of doxycycline post-exposure prophylaxis (dPEP) to reduce bacterial STIs among Kenyan women taking pre-exposure prophylaxis (PrEP). The overarching goal is to assess the effectiveness of dPEP on incidence of STIs while also balancing acceptability, cost, and impact on tetracycline resistance to inform public health policy. Participants will be randomized to receive dPEP and standard of care or the standard of care only. Questionnaires, focus group discussions, SMS, and in-depth interviews will be used to study acceptability and changes sexual behavior due to dPEP.

DETAILED DESCRIPTION:
This study is an open-label 1:1 randomized clinical trial of doxycyline PEP to reduce bacterial STIs - Neisseria gonorrhoeae, Chlamydia trachomatis, and T. pallidum (syphilis) - among Kenyan women taking PrEP. Participants will be counseled about the preliminary effectiveness data from IPERGAY, and the potential for resistance in STIs or other bacteria.

The primary study objectives are to 1) evaluate the effectiveness of doxycycline PEP (dPEP) to reduce STI infections in HIV-uninfected Kenyan women taking HIV PrEP; 2) assess the safety, tolerability, and acceptability of dPEP; 3)assess adherence to dPEP; 4) investigate the impact of dPEP on tetracycline resistance in N. gonorrhoeae and C. trachomatis; 5) measure the cost of dPEP and estimate the cost per case averted, budget impact, and affordability

Subjects will be randomized 1:1 to dPEP versus standard of care; randomization will be done in variable-sized blocks and using opaque envelopes opened at randomization. Participants assigned to dPEP will be instructed to take doxycycline 200 mg (two 100mg capsules) orally within 24 hours and up to 72 hours after each condomless sex act (consistent with IPERGAY) as frequently as daily if indicated but not more than once daily.

At Months 0,3,6 and 9, women randomized to dPEP will receive doxycycline, sufficient for up to daily use for 3 months (i.e., 180 capsules). Unused capsules will be counted at each quarterly follow-up visit and additional doxycycline will be provided. Participants will also be offered single- or multi-dose pill carriers for ease of dosing dPEP following exposures. All participants will receive quarterly visits for standard of care prevention services and collection of clinical and behavioral data, for a total of 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Age ≥18 years and ≤30 years old
* Female sex at birth
* HIV-seronegative at the time of last test within the past month and a current prescription for PrEP according to the national guidelines of Kenya (define PrEP eligibility as: partner of HIV-infected person not on ART or on ART for <6 months, >1 partner of unknown status, transactional sex, recent STI, recurrent HIV PEP use, inconsistent condom use, or injection drug use).

Exclusion Criteria:

* Pregnant
* Breastfeeding a child
* Allergy to tetracycline class
* Current medications which may impact doxycycline metabolism or that are contraindicated with doxycycline, as per the prescribing information. These include systemic retinoids, barbiturates, carbamazepine, phenytoin, and warfarin.
* Recent use of prolonged (more than 14 day course) antibiotics in the month prior to enrollment
* Active, clinically significant medical or psychiatric conditions that would interfere with study participation, at the discretion of the site investigator or designee.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 449 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baeten, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwach B, Kwena Z, Violette LR, Rono B, Odoyo JB, Oware K, Bukusi EA, Baeten JM, Mkandawire-Valhmu L, Stewart J; dPEP Kenya Study Team. Understanding barriers and facilitators to doxycycline post-exposure prophylaxis adherence among young women in western kenya: a qualitative study. BMC Infect Dis. 2025 Jul 1;25(1):855. doi: 10.1186/s12879-025-11209-6. PMID 40597823
- [Derived] Stewart J, Oware K, Donnell D, Violette LR, Odoyo J, Soge OO, Scoville CW, Omollo V, Mogaka FO, Sesay FA, McClelland RS, Spinelli M, Gandhi M, Bukusi EA, Baeten JM; dPEP Kenya Study Team. Doxycycline Prophylaxis to Prevent Sexually Transmitted Infections in Women. N Engl J Med. 2023 Dec 21;389(25):2331-2340. doi: 10.1056/NEJMoa2304007. PMID 38118022
- [Derived] Stewart J, Bukusi E, Sesay FA, Oware K, Donnell D, Soge OO, Celum C, Odoyo J, Kwena ZA, Scoville CW, Violette LR, Morrison S, Simoni J, McClelland RS, Barnabas R, Gandhi M, Baeten JM. Doxycycline post-exposure prophylaxis for prevention of sexually transmitted infections among Kenyan women using HIV pre-exposure prophylaxis: study protocol for an open-label randomized trial. Trials. 2022 Jun 16;23(1):495. doi: 10.1186/s13063-022-06458-8. PMID 35710444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | dPEP Intervention Arm | Standard of Care Arm
Started | 224 | 225
Completed | 220 | 222
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dPEP Intervention Arm | Standard of Care Arm | Total
Number analyzed (Participants) | 224 | 225 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 9 | 24
  Between 18 and 65 years | 209 | 216 | 425
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 24 [22 to 27] | 24 [22 to 27] | 24 [22 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 225 | 449
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African | 224 | 225 | 449
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 224 | 225 | 449

OUTCOME MEASURES:

1. Primary Outcome: Incidence of N. Gonorrhoeae, C. Trachomatis, or Early Syphilis Infection by Laboratory-based Diagnosis
Description: Combined incidence of N. gonorrhoeae, C. trachomatis, or early syphilis infection by by laboratory-based diagnosis (e.g., positive N. gonorrhoeae or C. trachomatis based on NAAT or syphilis based on four-fold increase in non-treponemal titers).
Time Frame: 12 months post enrolment
Population: Intention to treat, STI incidence events per 100 person-years
Measure: Number; unit: Events per 100 person-years
Arm/Group | dPEP Intervention Arm | Standard of Care Arm
Number analyzed (Participants) | 224 | 225
Events per 100 person-years | 25.1 | 29.0

ADVERSE EVENTS:
Time Frame: 12 months
Description: AEs, SAEs and social harms were recorded.
Arm/Group | dPEP Intervention Arm | Standard of Care Arm
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/225
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/225
Other Adverse Events (participants affected / at risk) | 40/224 | 12/225
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dPEP Intervention Arm (N=224) | Standard of Care Arm (N=225)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Social Harm (Social circumstances) | 4 (6) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Gastrointestinal Irritation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Lipoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 7 (8) | 7 (8)
Oral Yeast Infection (Infections and infestations) | 2 (2) | 0 (0)
Peptic Ulcers (Gastrointestinal disorders) | 2 (2) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Preterm Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Preterm Twin Cesarean Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (9) | 0 (0)
Achilles Tendon Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Hemorrhagic Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hyperemesis Gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Nuchal Cord (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Placental Abruption (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Renal Stones (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT04050540/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT04050540/SAP_001.pdf